CLINICAL TRIAL: NCT06976853
Title: Moving Beyond Inflammation as a Therapeutic Target for Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202504106
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide group (Experimental)
  Interventions: Drug: Tirzepatide
- Standard of Care Arm (Active Comparator)
  Interventions: Drug: Standard of care treatment

INTERVENTIONS:
Drug: Tirzepatide — Addition of tirzepatide to current biological therapy
  Arms: Tirzepatide group
Drug: Standard of care treatment — Intervention will be to change patient's current therapy to a 3rd or later advanced biologic patient have never been exposed to
  Arms: Standard of Care Arm

SUMMARY:
The purpose of this research study is to evaluate what type of treatment will be beneficial for people with Crohn's disease and difficult to treat inflammation in the small bowel. Current therapies are used to control the inflammation due to Crohn's disease in your digestive tract. In some patients, those therapies are not sufficient to fully treat the disease. This objective of this study is to evaluate the efficacy of a different type of therapy, tirzepatide, that may promote healing of the affected intestinal segment. To evaluate the efficacy of this medication, a member of the research team will ask patients questions about how they feel and observe whether this medication heals the their bowel at colonoscopy. A member of the research team will also use blood samples, stool samples and samples of the small intestine taken during a colonoscopy to understand how tirzepatide helps heal the intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 80 years of age, inclusive, at the time of consent
2. Confirmed diagnosis of Crohn's disease based on documented findings on endoscopy and histopathology
3. Active ileal or ileocolonic inflammation on colonoscopy defined as

   1. Ileal SES-CD > 4 with ulcer subscore > 1 (ulcers > 5mm)
4. Failure to respond to (primary or secondary non-response) at least 2 advanced class drugs, without evidence of immunogenicity (anti-TNFa only). Must have been at least 6 months optimized on most recent therapy without corticosteroids.

   1. Anti-TNF: Infliximab, Adalimumab, Certolizumab, Golimumab
   2. Anti-integrin agent: vedolizumab
   3. Anti-IL12/23 agent: Ustekinumab
   4. Anti-IL23: Risankizumab, Guselkumab, Mirikizumab
   5. JAK inhibitor: Upadacitinib
5. In post surgical patients, must be at least 6 months post-op with endoscopic evidence of ileal disease
6. In females: compliance to recommended birth control requirements

Exclusion Criteria:

1. Age < 18 or > 80 years
2. Pregnant or Breastfeeding female
3. Diagnosis of ulcerative colitis, indeterminate colitis, microscopic colitis, ischemic colitis, radiation colitis, diverticular disease-associated colitis, toxic megacolon, active infectious colitis or positive test for Clostridioides Difficile toxin at screening
4. BMI < 25
5. Current or previous diagnosis of anorexia nervosa
6. Type 1 or Type 2 diabetes
7. Use of concomitant hypoglycemic agents
8. Personal or family history of medullary thyroid carcinoma
9. History of multiple endocrine neoplasia
10. Known serious hypersensitivity to tirzepatide or any of its excipients
11. Have functional or post-operative short-bowel syndrome
12. Had intestinal resection ≤ 24 weeks prior to inclusion or other intra-abdominal surgeries ≤ 12 weeks prior to study inclusion
13. Active treatment with steroids*
14. Positive stool test for parasites, C. Diff or stool culture for pathologic bacteria within 30 days prior to enrollment
15. Current stricture not passable with an endoscope
16. Impending need for surgery per investigator
17. Have an ileostomy or a colostomy
18. In females: refusal to comply to recommended birth control requirements *Corticosteroids have metabolic and hormonal effects which we are concerned may interfere with study outcomes and metabolic changes in the population. This exclusion criteria will allow the study population to be standardized across all patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion and number of participants who have treatment emergent adverse events, serious adverse events, discontinuation of study intervention due to adverse events and injection-site reactions by CTCAE v4.0 | From enrollment to the end of treatment at month 7
Number of participants who achieve various doses of Tirzepatide at increments of 2.5 mg, up to 15 mg | From enrollment to the end of treatment at month 7
Proportion and number of participants with endoscopic remission as defined by SES-CD < 4 with no ulcer subscore >1. | From enrollment to the end of treatment at month 7

SECONDARY OUTCOMES:
Proportion and number of participants with endoscopic response as defined by (↓SES-CD 50%) | From enrollment to the end of treatment at month 7
Proportion and number of participants who achieve clinical remission/response defined by Crohn's disease activity index < 150 for clinical remission or a decrease from baseline by at least 100 points on CDAI | From enrollment to the end of treatment at month 7
Proportion and number of participants who achieve clinical remission defined by a Harvey Bradshaw Index < 5 | From enrollment to the end of treatment at month 7
Proportion and number of participants who achieve improvement from baseline in the Short Inflammatory Bowel Disease Quality of Life Questionnaire in four domains, bowel symptoms, emotional health, systemic systems and social function. Questions are score | From enrollment to the end of treatment at month 7
Proportion and number of participants who achieve improvement from baseline in visceral adipose tissue, the total body fat percentage, fat mass index by DEXA | From enrollment to the end of treatment at month 7
Rates of remission in each group (3rd advanced therapy, tirzepatide 5mg dosing, tirzepatide escalated dosing) | From enrollment to the end of treatment at month 7

CONTACTS AND LOCATIONS:
Overall Officials: Parakkal Deepak, MBBS, MS, Principal Investigator — Washington University School of Medicine GI Division; Louis Cohen, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Andres Yarur, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York